CLINICAL TRIAL: NCT02424474
Title: Fetal Aneuploidies Screening (21,18 and 13) by Cell Free Fetal DNA Analysis. Pilot Study in Low Risk Population and Pregnant Women After in Vitro Fertilisation (IFV)
Brief Title: T21,18 and 13 Screening by Cell Free Fetal DNA in Low Risk Patients
Acronym: DEPOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P141001
Record Dates: First submitted 2015-04-08; First posted 2015-04-23 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2016-09

CONDITIONS: Trisomy 21, 18 and 13 Screening
Keywords: cell free fetal DNA; general population; screening; trisomy 21; IVF
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genetic NIPT and regular serum screening (Experimental): All woman will be tested using the two tests, genetic NIPT (Non Invasive Prenatal Testing) and regular serum screening.
  Interventions: Device: Genetic NIPT; Biological: Regular serum screening

INTERVENTIONS:
Device: Genetic NIPT — Both tests are realized in a population of pregnant women (with and without in vitro fertilisation (IVF)) concomitantly at the same time.
Biological: Regular serum screening
  Other Names: Usual screening

SUMMARY:
The purpose of this study is to evaluate the performance of non invasive screening in a population of pregnant women with and without in vitro fertilisation (IVF) concomitantly to regular first trimester trisomy 21 (T21) screening using maternal age, nucal fold measurement and serum screening.

DETAILED DESCRIPTION:
All pregnant women in 9 institutions in France will be offer both regular first trimester screening for trisomy 21 (T21) and cell free DNA non invasive (NI) screening test at the same time. Specificity and the positive and negative predictive values of the NI test will be analysed. The population will be divided in women who did and did not get pregnant after an In vitro fertilisation (IVF) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Singleton pregnancy
* Having a spontaneous pregnancy or obtained by AMP ,
* Having chosen to carry out a screening of the T21 to the first or second trimester of pregnancy ,
* Gestational age >=10 weeks of amenorrhea
* Consenting to invasive prenatal diagnosis,
* Having health insurance,
* Having signed the informed consent

Exclusion Criteria:

* The Patients whose fetus has an abnormality on the first trimester ultrasound including nuchal translucency > 3.5mm ,
* Participant to another biomedical research.
* Pregnancy twins including the presence of a twin vanishing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance measured by specificity (%) of genetic Non Invasive Prenatal Testing (NIPT) in the two populations (with and without IVF) compared to regular serum screening | Between the 11th and the 13th week of amenorrhea

SECONDARY OUTCOMES:
Diagnostic performance measured by positive predictive values (%) of genetic NIPT (Non Invasive Prenatal Testing) in the two populations compared to regular serum screening | Between the 11th and the 13th week of amenorrhea
  positive ad negative predictive values of NIPT in the two populations of woman with and without IVF.
Diagnostic performance measured by negative predictive values (%) of genetic NIPT (Non Invasive Prenatal Testing) in the two populations compared to regular serum screening | Between the 11th and the 13th week of amenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Benachi, MD, PhDi, Principal Investigator — AP-HP, Antoine Béclère Hospital
Locations (1):
- AP-HP, Antoine Béclère Hospital, Clamart, France

REFERENCES:
- [Derived] Dabi Y, Guterman S, Jani JC, Letourneau A, Demain A, Kleinfinger P, Lohmann L, Costa JM, Benachi A. Autoimmune disorders but not heparin are associated with cell-free fetal DNA test failure. J Transl Med. 2018 Dec 3;16(1):335. doi: 10.1186/s12967-018-1705-2. PMID 30509296
- [Derived] Costa JM, Letourneau A, Favre R, Bidat L, Belaisch-Allart J, Jouannic JM, Quarello E, Senat MV, Broussin B, Tsatsaris V, Demain A, Kleinfinger P, Lohmann L, Agostini H, Bouyer J, Benachi A. Cell-free fetal DNA versus maternal serum screening for trisomy 21 in pregnant women with and without assisted reproduction technology: a prospective interventional study. Genet Med. 2018 Nov;20(11):1346-1353. doi: 10.1038/gim.2018.4. Epub 2018 Mar 1. PMID 29493578